CLINICAL TRIAL: NCT00840697
Title: Facilitating and Inhibiting Factors and Effect of Interventions in Return to Work for Patients With Neck and Low Back Pain
Brief Title: Effect of Interventions in Return to Work for Patients With Neck and Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Professor, PhD, Erik bautz-Holter, Ullevaal University Hospital, 0407 Oslo, Norway
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: return to work and exercise
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-05

CONDITIONS: Low Back Pain; Neck Pain
Keywords: low back pain; neck pain; return to work; exercises; cognitive intervention
MeSH Terms: conditions — Low Back Pain; Neck Pain; Motor Activity | interventions — Exercise; Return to Work; Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Work related rehabilitation (Active Comparator): work related rehabilitation and exercises
  The workplace intervention includes two steps:
  Evaluations of the work site: The occupational ergonomists task is to identify conditions at the work site, as for instance ergonomic, work demand and relations to the employer and colleagues.
  Therapeutic Return to work: The occupational ergonomists will organize contacts and meetings between the employer and the patients and make a schedule for return to work. The therapeutic return-to-work-process will take place at the work place, with progressively more days at work and progressively increasing tasks.
  Exercises comprises of treatment in groups. The treatment includes exercises, both strength and fitness, in addition to cognitive intervention of how to manage pain and work.
  Interventions: Behavioral: Exercises and work related rehabilitation
- Brief intervention (Active Comparator): 1 consultation at the physiotherapist, which give advise and a summary talk with the physician
  Interventions: Behavioral: Brief intervention
- Multidisciplinary exercise group (Active Comparator): 10 days of exercise and cognitive treatment group
  Interventions: Behavioral: multidisciplinary exercise group

INTERVENTIONS:
Behavioral: Exercises and work related rehabilitation — Treatment in groups, twice a week for 3 weeks. The treatment includes exercises, cognitive intervention and work related rehabilitation. The exercises include fitness, strength and stretching
  Other Names: return to work; Low back pain; Behavioral
  Arms: Work related rehabilitation
Behavioral: Brief intervention — 1 consultation at the physiotherapist, which give advice Summary talk with the physician about activity and work when having neck- and low back pain
  Arms: Brief intervention
Behavioral: multidisciplinary exercise group — 10 days during 3 weeks. Treatment in groups, exercise and cognitive treatment
  Arms: Multidisciplinary exercise group

SUMMARY:
Low back pain is a usual condition in the western countries and several treatments available for patients with "non-specific low back pain". According to the European guidelines both Brief intervention and exercise/cognitive intervention are effective treatments with regard to pain and function (www.backpaineurope.org), but none have documented effect on return to work.

The challenges for health personnel is not cure of the patients back pain, but to build up rehabilitation programs which focus on disability and work incapacity, in patients which are at risk of loosing their work. Dr. P. Loisel, Montreal, Canada", has since 1995 treated patients with back pain according to the "The PREVICAP model - (PREVention of work handICAP)", where the main purpose with work-related program is to prevent prolonged disability and to help patients back to work. Loisel demonstrated that the PREVICAP models accelerated the "return to work" factor by a factor 2.4 (p=0.01). The PREVICAP model had also been evaluated in Amsterdam, by Dr. Anema with the same results.

At the Back Clinic, Ullevål University Hospital we are presently involved in a randomized controlled trial after the PREVICAP model, where patients are randomized to Brief intervention including a work-related intervention or usual care. All included patients in both groups, will have a clinical examination by specialist in Physical Medicine and Rehabilitation and advice from a physiotherapist. The current study replaces Brief intervention with an exercise - and a work-related program, so patients with non-specific LBP will be randomized to an exercise and work-related program or usual care.

The main purpose of this study

* to investigate if rehabilitation programs specifically focusing on the return to work process will reduce sickness absence and disability pension in patients with neck and low back pain.
* to assess the work-, individual- and health factors and their interrelationship predicting sickness absence and work disability.
* to compare results from the rehabilitation program with results from rehabilitation program in Toronto
* to which extent are the patients met by actions from employers and employment services, and does is influence sickness absence and disability.
* do these actions represent favourable cost benefit for the work places and the society

DETAILED DESCRIPTION:
Background:

Norway has the highest sickness absence of the Scandinavian countries, with a cost of about 40 milliard kr each year. In addition about 500 000 receive rehabilitation or disability pension comprising a cost of 75 milliard kr. Musculoskeletal pain is the most common cause of sickness absence and among the 3 most common causes of disability pension in Norway [1]. For young subjects (<40 years) musculoskeletal disorders also represent the most common cause for disability pension [2]. Neck and low back pain comprise the majority of patients with musculoskeletal disorders. Hence, several actions have been initiated in order to reduce sickness absence and improve participation in the working life.

The agreement about "including work life" ("IA avtalen") was introduced in 2001, and represented a joint effort from the government, the employers' organizations and the labor organizations. The superior aim was to prevent sickness absence and promote the inclusion in the working life despite sickness and disability. However, it soon became clear that there was a contradiction between the goals of reducing sickness absence and including subjects with diseases and disabilities. In addition it became clear that the knowledge about the factors facilitating participation in working life was scarce. Groups with low education level, foreign origin, women and subjects with chronic diseases dominating the sickness absence statistics were not reached [3], and effective strategies to improve also these groups employment were sought. Hence, a committee leaded by the prime minister granted above 600 mill kr in order to reduce the sickness absence about 2.5 %. The committee recognized the need of reinforcing the collaboration between the employers and the employed. However, the main focus the need of a coordinated effort from the health care system and the social security and employment service. The latter two are fused to one organisation in Norway termed "NAV" (Nye arbeids og velferds etaten). Necessary health services need to be provided immediately and a close collaboration with the social security and employment service as well as the employers.

Most of the patients with neck and low back pain have benign and self-limited conditions, which they nevertheless experience as pain full and disabling [4;5]. According to the European guidelines, exercise and cognitive intervention has good effects on pain and function for patients with low back pain [6] (www.backpaineurope.org). Multimodal treatment including exercises has also been shown effective for patients with neck pain [7]. However, these treatment modalities do not seem sufficiently effective in order to improve return to work [8].

Neck and low back pain is a multifactorial problem, which is not only due to workers' medical characteristics, but is also closely related to environmental factors, such as the workplace and individual factors. Physical factors like heavy lifting, vibration and posture demands may be of importance for low back pain [9;10]. The working life of today demanding increasingly use of computers is a risk factor for neck, shoulder and arm disorders. Particularly, where the work station is poorly designed and the duration of the computer use above 4 hours a day there is a risk for pain development [10]. Even more important is the psychosocial environment at work. Factors such as control over the work situation, demands and support from the colleagues and leader are of importance [11]. The compensation system and the interaction between all stakeholders in the disability problem and the health care system are of importance for the return to work [12;13]. In addition time is a significant factor, with reduced return to work after longer periods of sick leave [14]. Among the individual factors of major importance is educational level [15], which of course is related to socioeconomic class. Age, gender and cultural background are also well known predictors for sickness absence and disability pension [16], which adds to the higher prevalence of musculoskeletal pain in these groups [17]. Interventions at the work place coordinated with early contact with worker by workplace, contact between healthcare provider and workplace has also been shown to improve return to work [18].

Thus, return to work is not dependent on one single step, but a challenging process where the patient, health professionals, employers and employment system must interact. A particular challenge is to build up rehabilitation-programs for patients at risk of loosing their work [19]. Dr. P. Loisel, Montreal, Canada" [20], have since 1995 treated patients with low back pain according to the "The PREVICAP modell - (PREVention of work handICAP)". The main purpose with work-related program is to prevent prolonged disability and helping patients to return to work. This process includes identification of factors on the workplace which contribute to the absence of work. These factors include physical, ergonomic, psychosocial, interpersonal conflicts and administrative problems. Subsequently "workplace intervention" is initiated. This is a rehabilitation-program centered at the workplace, allowing a graded transition from the clinical setting to the workplace. Parallel with the workplace intervention the patients enter into a short exercise-program, adjusted to the workplace intervention. The Previcap models have been evaluated in randomized controlled trials and accelerated the return to work by a factor 2.4 and the most important effect came from the workplace intervention, which accelerated the return to work with a factor 1.9. Patients randomized to the Previcap model had 60 days absence from work, compared to 120 days in the control group [20;21]. The Previcap-model have also been evaluated in Amsterdam, by Dr. Anema and he demonstrated a significant difference in the return to work rate between patients randomized to "Workplace intervention" and to usual treatment. This type of interventions has not been tried on patients with neck pain, and in general the knowledge regarding neck pain is poorer than for low back pain. Hence, Sconstein et al [8] performing a Cochrane review, concluded that there is an urgent need for well designed randomised studies trying to facilitate return to work in patients with neck pain.

It is also important to take into account that the predictors for sickness absence are different from the factors determining return to work [22]. This is largely embezzled in the intervention strategies. Another shortcoming is failure to meet the needs of the employees with disabilities [23]. That may be chronic back conditions that cannot be cured, or the combined cause of back pain and comorbidity which is frequent in this population [24]. This is particularly important as employment seems to be a very important factor for mental health in subjects with disabilities [25]. Research focusing on the interrelationship between these different factors is lacking. This type of knowledge is needed in order to improve the intervention strategies. It is also obvious that success can only be achieved if the employment services and stakeholders contribute. Hence, the research in this field calls for a joint effort between the health care services, employers and employment services.

At Ulleval University Hospital (UUH) and at St Olavs hospital the health care for patients with neck-and back pain has been organised in multi-professional units, taking care of a about 4000 and 2000? patients, respectively, at an annual basis. Within this system it is possible to provide necessary diagnostic evaluation and medical treatment. The ongoing NAV projects at both institutions provide the possibility to offer medical care within 2 weeks. Multimodal treatments including exercises are also provided. At UUS, the PREVICAP model is implemented and evaluated against usual treatment for patients with low back pain in a randomized trial. However, patients with neck pain are not included. Hence, a main intention is to evaluate the PREVICAP model in a randomized trial including patients with neck pain. In a worker population the psychosocial factors at work including relationship between demand and control [26] as well as the balance between effort and rewards [27] are shown to be of importance. Such a comprehensive assessment of patient reported work-related factors has not previously been performed in the specialized health care. These factors will be combined with the medical assessment and personal factors in the multiple prediction models, in order to single out combinations of factors of importance.

Although, The PREVICAP model had shown good results on Return to work, in Montreal, and Amsterdam, it is unknown how this model will work out in other countries, due to differences in culture, working terms and compensatory system? So, we will collaborate with the research group in Toronto (D.Cassidy, Health Network Rehabilitation Solutions,Toronto Western Hospital) to up multinational studies for Return to work-Rehabilitation for patients with neck and back complaints.

The process of returning to work can only be completed when the identified problems can be met with adequate actions at the work place and NAV. These actions also reduce costs associated with work disability duration [18;28]. Few studies have addressed how the collaboration between the health care system and both employers and employment services. Hence, to which extent the advised adaptations at the work place are taken care of as well as the support given by NAV need to be assessed and related to the outcome of participation in working life. And at last, the costs and potential socioeconomic consequences of these actions need to be assessed.

The main purpose of this study is to combine the knowledge of the medical aspect of neck-and back pain with the knowledge of organizational and compensatory structure, occupational- and socioeconomic factors for investigating these factors influence and cause of the phenomenon sick-leave.

The specific aims are:

* to assess the work-, individual- and health factors and their interrelationship predicting sickness absence and work disability.
* to investigate if rehabilitation programs specifically focusing on the return to work process will reduce sickness absence and disability pension in patients with neck and low back pain.
* to compare results from the rehabilitation program with results from rehabilitations program in Toronto
* to which extent are the patients met by actions from employers and employment services, and does is influence sickness absence and disability.
* do these actions represent favorable cost benefit for the work places and the society

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain, sick listed for less than 1 year and who are permanently employed

Exclusion Criteria:

* Patients with infection, tumors, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome, spinal stenosis or spondylolysis/listesis, serious somatic disease and/or psychic disease and patients with with poor proficiency in Norwegian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
return to work rate | week

SECONDARY OUTCOMES:
Cost benefit, predictors (work, individual and health factors) of poor return to work rate, | year

CONTACTS AND LOCATIONS:
Overall Officials: Erik Bautz-Holter, Professor, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Marchand GH, Myhre K, Leivseth G, Sandvik L, Lau B, Bautz-Holter E, Roe C. Change in pain, disability and influence of fear-avoidance in a work-focused intervention on neck and back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2015 Apr 21;16:94. doi: 10.1186/s12891-015-0553-y. PMID 25896785